CLINICAL TRIAL: NCT00422747
Title: Early Diagnosis of Asthma in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Netherlands Asthma Foundation (Other); Stichting Astma Bestrijding, The Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL17407.000.07/2007-001817-40
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: asthma; transient wheezing; early diagnosis; exhaled air; nitrogen monoxide; airway resistance
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- beclomethasondipropionate (Experimental): 2 x 100 ug dd for two months, via aerochamber
  Interventions: Drug: beclomethasondipropionate

INTERVENTIONS:
Drug: beclomethasondipropionate — 2 x 100 ug dd for two months, via aerochamber
  Other Names: Qvar Extra Fijn

SUMMARY:
The overall aim of the study is an early asthma diagnosis in young children by the use of non-invasive biomarkers of airway inflammation /oxidative stress in exhaled air, and early lung function measurements

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-3 years, with recurrent respiratory symptoms suggestive of asthma
* Children aged 2-3 years, with no or minor respiratory symptoms

Exclusion Criteria:

* Mental retardation
* Cardiac anomalies
* Congenital malformations
* Other diseases of the lungs/airways
* Chronic systemic inflammatory diseases like M. Crohn
* The inability to perform lung function measurements and/or exhaled air collection

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2007-04; Primary Completion 2011-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
- definite asthma diagnosis - biomarkers in exhaled breath | 6 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Edward Dompeling, PhD MD, Principal Investigator — Dept. of Paediatric Pulmonology, Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Klaassen EM, van de Kant KD, Jobsis Q, van Schayck OC, Smolinska A, Dallinga JW, van Schooten FJ, den Hartog GJ, de Jongste JC, Rijkers GT, Dompeling E. Exhaled biomarkers and gene expression at preschool age improve asthma prediction at 6 years of age. Am J Respir Crit Care Med. 2015 Jan 15;191(2):201-7. doi: 10.1164/rccm.201408-1537OC. PMID 25474185
- [Derived] van de Kant KD, van Berkel JJ, Jobsis Q, Lima Passos V, Klaassen EM, van der Sande L, van Schayck OC, de Jongste JC, van Schooten FJ, Derks E, Dompeling E, Dallinga JW. Exhaled breath profiling in diagnosing wheezy preschool children. Eur Respir J. 2013 Jan;41(1):183-8. doi: 10.1183/09031936.00122411. PMID 23277518
- [Derived] van de Kant KD, Koers K, Rijkers GT, Lima Passos V, Klaassen EM, Mommers M, Dagnelie PC, van Schayck CP, Dompeling E, Jobsis Q. Can exhaled inflammatory markers predict a steroid response in wheezing preschool children? Clin Exp Allergy. 2011 Aug;41(8):1076-83. doi: 10.1111/j.1365-2222.2011.03774.x. Epub 2011 May 30. PMID 21623968
- [Derived] van de Kant KD, Klaassen EM, Jobsis Q, Nijhuis AJ, van Schayck OC, Dompeling E. Early diagnosis of asthma in young children by using non-invasive biomarkers of airway inflammation and early lung function measurements: study protocol of a case-control study. BMC Public Health. 2009 Jun 29;9:210. doi: 10.1186/1471-2458-9-210. PMID 19563637